CLINICAL TRIAL: NCT00907894
Title: A Phase I, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of Telbivudine (LDT600) in Children and Adolescents With Chronic Hepatitis B
Brief Title: Pharmacokinetics and Safety of Single-Dose Telbivudine in Children and Adolescents With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLDT600A2104; EudraCT 2007-006218-40
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-09

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B,; telbivudine,; pharmacokinetics,; safety,; tolerability,; pediatric
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

ARMS (3):
- Stratum 1 (Experimental)
  Interventions: Drug: LDT600 (Telbivudine)
- Stratum 2 (Experimental)
  Interventions: Drug: LDT600 (Telbivudine)
- Stratum 3 (Experimental)
  Interventions: Drug: LDT600 (Telbivudine)

INTERVENTIONS:
Drug: LDT600 (Telbivudine) — LDT600 (Telbivudine)

SUMMARY:
This is a Phase I, open-label, single-dose study to evaluate the pharmacokinetics and safety of LDT600 in pediatric and adolescent patients with chronic hepatitis B infection.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents patients
* HBsAg seropositive

Exclusion criteria:

* Decompensated liver disease (Child-Turcotte-Pugh (CTP) Score≥7, Class B and C)
* Prior anti-HBV therapy within 30 days of study drug dosing.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
LDT600 plasma concentration and pharmacokinetic (PK) parameters of exposure (Cmax and AUC) | 6 days
  To evaluate the single-dose pharmacokinetics of LDT600 in pediatric and adolescent patients (2-18 years of age) with chronic hepatitis B (CHB) infection.

SECONDARY OUTCOMES:
Safety assessments will include vital signs, ECG and incidence of adverse events and serious adverse events. | 6 days
  To evaluate the safety and tolerability of LDT600 in pediatric and adolescent patients with chronic hepatitis B infection

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Brussels, Belgium
- Germany (3):
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigator Site, Starnberg
  - Novartis Investigator Site, Wuppertal
- Philippines (2):
  - Novartis Investigator Site, Manila
  - Novartis Investigator Site, Quezon City
- Novartis Investigator Site, Birmingham, United Kingdom

REFERENCES:
- [Derived] Stein DS, Ke J, Uy G, Bosheva M, Qi Y, Praestgaard J; LDT600A2104 Study Team. Phase I, open-label, single-dose study to evaluate the pharmacokinetics and safety of telbivudine in children and adolescents with chronic hepatitis B. Antimicrob Agents Chemother. 2013 Sep;57(9):4128-33. doi: 10.1128/AAC.00117-13. Epub 2013 Jun 17. PMID 23774433
- See also: Results for CLDT600A2104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7003